CLINICAL TRIAL: NCT02984462
Title: Is Fixation of Percutaneous Akin Osteotomy Enhanced First Ray Post-operative Mobility? A Prospective Randomized Study.
Brief Title: Akin Osteotomy With or Without Fixation
Acronym: AKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2015/39
Record Dates: First submitted 2016-10-27; First posted 2016-12-07 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Hallux Valgus
Keywords: percutaneous; non-fixed; Akin ;; osteotomy
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- screw fixation (Experimental): Surgical Percutaneous Akin osteotomy with fixation by a percutaneous cannulated screw and forefoot surgery dressing.
  Interventions: Procedure: percutaneous Akin osteotomy
- No fixation (No Intervention): Surgical Percutaneous Akin osteotomy non-fixed, hold by forefoot surgery dressing.

INTERVENTIONS:
Procedure: percutaneous Akin osteotomy — The act to AKIN is osteotomy in percutaneous; This technique can be performed with or without fixation, and both methods make reference in the literature. With fixation method to get rid of the risk of loss of the surgical reduction of the misalignment, but requires an additional surgical procedure marked by the implementation of a percutaneous cannulated screw on part of the osteotomy. Without fixing method allows to get rid of this gesture, and risk a possible annoys by osteo-synthesis material. Surgical dressings of surgery of hallux valgus allow to keep the reduction for 15 days. Both techniques give excellent results and are performed in our service of routinely.
  Arms: screw fixation

SUMMARY:
The study is a prospective randomized study about hallux valgus surgery. The investigator try to assess if the fixation of percutaneous Akin osteotomy with a cannulated screw have an incidence in the first ray mobility since the two technics ( fixation and no-fixation) are described and practiced, and since the stiffness of the first metatarso-phalangeal joint is determinant in the result of this functional surgery.

DETAILED DESCRIPTION:
It's a prospective monocentric randomized work about forefoot surgery. Every patient included undergoes an hallux valgus chevron osteotomy of the first metatarsal associated with a percutaneous Akin osteotomy of the first phalange. The investigators study the impact of the fixation of percutaneous Akin osteotomy ( osteotomy of the first phalange of hallux) with two arms: one with fixation of the percutaneous Akin osteotomy, and one with a non-fixed percutaneous Akin osteotomy This study as been approved by Institutional review board; written informed consent is required for all patients before inclusion.

The clinic follow-up of each patients included in the study will be the same of the normal follow-up for this type of surgery in our practice. This includes clinical exam, radiologic exam, and functional score AOFAS before surgery, at 6 weeks after the surgery, four months after surgery and finally one year after the surgery.

The primary outcome measure which is the first metatarso-phalangeal global mobility will be blindly measure by an observator.

ELIGIBILITY:
Inclusion Criteria:

* patient which need hallux valgus surgery

Exclusion Criteria:

* hallux rigidus
* Trouble of rotation of the the hallux
* Rheumatoid forefoot
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Global Mobility in degrees of the metatarso-phalangeal joint of the hallux one year after the surgery. | 12 months

SECONDARY OUTCOMES:
Angle between Metatarsus 1 and Phalanx 1 | 12 months
Angle between Metatarsus 1 and Metatarsus 2 | 12 months
Angle between Phalanx 1 and Phalanx 2 | 12 months
Distal Metatarsal Articular Angle | 12 months
DM2A angle, calculated preoperatively by measuring the angle between the metatarsal diaphysis M2 and the tangent at the vertex of the distal articular surface | 12 months
DM2A angle, calculated at last follow-up by measuring the angle between the metatarsal diaphysis M2 and the tangent at the vertex of the distal articular surface | 12 months
Kitaoka Score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien LUCAS Y HERNADEZ, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique; University Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux - Hospital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No